CLINICAL TRIAL: NCT01640353
Title: Sacroiliac Joint Fusion With iFuse Implant System (SIFI)
Acronym: SIFI
Status: Completed | Type: Observational
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 300101
Record Dates: First submitted 2012-07-06; First posted 2012-07-13 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Degenerative Sacroiliitis; Sacroiliac Joint Disruption
Keywords: si joint; si joint pain; si joint injury; si joint treatment; si joint injections; si joint inflammation; si joint problems; si joint symptoms; hypermobile si joint; si joint arthritis; si joint pain treatment; inflamed si joint; si joint sclerosis; locked si joint; si joint injuries; si joint disease; si joint infection; sacroiliac joint pelvic pain; sacroiliac joint arthritis treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the use of the iFuse Implant System to treat degenerative sacroiliitis (arthritis of the SI joint) and sacroiliac disruption (abnormal separation or tearing of the sacroiliac joint). The iFuse Implant System (iFuse device) is a medical device that is surgically implanted into the sacroiliac (SI) joint during a minimally invasive surgical procedure (one that uses a smaller incision and less damage to the skin and other tissues than standard surgery). The purpose of implanting the device is to stabilize and fuse the SI joint.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-70 at time of screening

2. Patient has lower back pain for >6 months inadequately responsive to conservative care

3. Diagnosis of sacroiliac joint disruption or degenerative sacroiliitis based on ALL of the following:

1. Patient has pain at or close to the posterior superior iliac spine (PSIS) with possible radiation into buttocks, posterior thigh or groin and can point with a single finger to the location of pain (Fortin Finger Test), and
2. Patient has at least 3 of 5 physical examination maneuvers specific for the SI joint (see Table 3), and
3. Patient has improvement in lower back pain numeric rating scale (NRS) of at least 50% after injection of local anesthetic into affected SI joint(s) (see Section 3.6.4), and
4. One or more of the following:

i. SI joint disruption:

1. Asymmetric SI joint widening on X-ray or CT scan
2. Leakage of contrast on diagnostic arthrography

ii. Degenerative sacroiliitis:

1. Radiographic evidence of SI joint degeneration, including sclerosis,osteophytes, subchondral cysts, or vacuum phenomenon on CT or plain film, or
2. Due to prior lumbosacral spine fusion

4. Baseline Oswestry Disability Index (ODI) score of at least 30% 5. Baseline SI joint pain score of at least 50 on 0-100 mm visual analog scale 6. Patient has signed study-specific informed consent form 7. Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements

Exclusion Criteria:

1. Severe back pain due to other causes, such as lumbar disc degeneration, lumbar disc herniation, lumbar spondylolisthesis, lumbar spinal stenosis, lumbar facet degeneration, and lumbar vertebral body fracture
2. Other known sacroiliac pathology such as:

   1. Sacral dysplasia
   2. Inflammatory sacroiliitis (e.g., ankylosing spondylitis or other HLA-associated spondyloarthropathy)
   3. Tumor
   4. Infection
   5. Acute fracture
   6. Crystal arthropathy
3. History of recent (< 1 year) major trauma to pelvis
4. Previously diagnosed osteoporosis (defined as prior T-score <-2.5 or history of osteoporotic fracture).
5. Osteomalacia or other metabolic bone disease
6. Chronic rheumatologic condition (e.g., rheumatoid arthritis)
7. Any condition or anatomy that makes treatment with the iFuse Implant System infeasible
8. Chondropathy
9. Known allergy to titanium or titanium alloys
10. Use of medications known to have detrimental effects on bone quality and soft-tissue healing
11. Prominent neurologic condition that would interfere with physical therapy
12. Current local or systemic infection that raises the risk of surgery
13. Patient currently receiving or seeking worker's compensation, disability remuneration, and/or involved in injury litigation.
14. Currently pregnant or planning pregnancy in the next 2 years
15. Patient is a prisoner or a ward of the state.
16. Known or suspected drug or alcohol abuse
17. Diagnosed psychiatric disease (e.g., schizophrenia, major depression, personality disorders) that could interfere with study participation
18. Patient is participating in an investigational study or has been involved in an investigational study within 3 months prior to evaluation for participation

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with SI joint pain due to degeneration or disruption of the SI joint
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Duhon, MD, Principal Investigator — University of Colorado, Denver
Locations (26):
- United States (26):
  - Spine and Neuro Center, Huntsville, Alabama
  - Silicon Valley Spine, Campbell, California
  - BASIC Spine, Newport Beach, California
  - Southern California Center for Neuroscience and Spine (SCCNS), Pomona, California
  - St. Mary's Spine, San Francisco, California
  - Neurosurgical and Spine Specialists, Parker, Colorado
  - Orthopaedic Clinic of Daytona Beach, Daytona Beach, Florida
  - The Orthopaedic Institute/NFRMC, Gainsville, Florida
  - Bartow Regional Medical Center, Lakeland, Florida
  - Piedmont Orhopaedics, Macon, Georgia
  - Orthopaedic Center of Southern Illinois, Mount Vernon, Illinois
  - Bluegrass Orthopaedics & Hand Care Research, Lexington, Kentucky
  - Columbia Orthopaedic Group, Columbia, Missouri
  - Midwest Division-RMC, LLC,-Research Medical Center, Kansas City, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - Alice Peck Day Memorial Hospital, Lebanon, New Hampshire
  - Manhattan Orthopedic Spine, PLLC, New York, New York
  - Orthopedic and Reconstructive Center (formally)Health Research Institute, Oklahoma City, Oklahoma
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - East Tennesse Brain & Spine Center, Johnson City, Tennessee
  - Brazos Spine, College Station, Texas
  - Texas Back Institute, Plano, Texas
  - Precision Spine Care, Tyler, Texas
  - Virginia Spine Institute, Reston, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data is shared with YODA project.

REFERENCES:
- [Derived] Dat KO, Cher D, Polly DW. Effects of BMI on SI joint fusion outcomes: examining the evidence to improve insurance guidelines. Spine J. 2024 May;24(5):783-790. doi: 10.1016/j.spinee.2023.11.015. Epub 2023 Dec 9. PMID 38081463

RESULTS

PARTICIPANT FLOW:
Groups:
- Sacroiliac Joint Fusion: SI Joint Fusion with iFuse implant system
Period: Overall Study
Arm/Group | Sacroiliac Joint Fusion
Started | 194
Treated | 172
Month 1 | 171
Month 3 | 169
Month 6 | 168
Month 12 | 160
Month 18 | 150
Completed | 149
Not Completed | 45
Not completed — Withdrew prior to treatment | 10
Not completed — Withdrawn from analysis at term site | 12
Not completed — Withdrawal by Subject | 5
Not completed — Death | 2
Not completed — Early site termination | 3
Not completed — Lost to Follow-up | 12
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sacroiliac Joint Fusion
Number analyzed (Participants) | 172
Age, Continuous [Mean (Full Range); unit: Years] | 50.9 [23.5 to 71.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 165
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 166
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 172
Baseline SIJ pain [Mean (Standard Deviation); unit: units on a scale] — The Visual Analog Scale (VAS) is a 100 mm line on which the subjects mark their pain rating. 0= no pain and 100= worst pain imaginable.
  units on a scale | 79.8 (12.8)
Baseline ODI [Mean (Standard Deviation); unit: units on a scale] — Oswestry Disability Index is a validated measure of disability related to low back pain. There are 10 sections, each with a score between 0-5. If all sections are answered, the total possible score is 50/50 = 100% which is the worst disability possible on the scale. (0/50 = no disability at all.) If any section is skipped by the study participant, the total possible score for that section is removed from the denominator. Example - section 8 skipped, total possible score is 45/45 = 100%.
  units on a scale | 55.2 (11.5)
Baseline EQ-5D [Mean (Standard Deviation); unit: units on a scale] — EuroQoL-5D (EQ-5D) is a standardized instrument to measure health state. It is a single index value for health status. A score of 0 would = worst imaginable health state while a score of 1.0 would be best imaginable health state.
  units on a scale | .43 (0.18)
Baseline SF-36 PCS [Mean (Standard Deviation); unit: units on a scale] — The Short Form 36 health survey (SF-36) is a 36-item patient reported health questionnaire to measure quality of life across 8 domains. The PCS is the Physical Component Summary score. 0% would represent the lowest or worst possible level of functioning while 100% would represent the highest / best possible level of functioning.
  units on a scale | 31.7 (5.6)
SF-36 MCS [Mean (Standard Deviation); unit: units on a scale] — The Short Form 36 health survey (SF-36) is a 36-item patient reported health questionnaire to measure quality of life across 8 domains. The MCS is the Mental Component Summary score. 0% would represent the lowest or worst possible level of functioning while 100% would represent the highest / best possible level of functioning.
  units on a scale | 38.5 (11.3)
Duration of prior pain [Mean (Full Range); unit: Years] | 5.1 [0.43 to 41.08]

OUTCOME MEASURES:

1. Primary Outcome: Subject Success
Description: Composite endpoint of reduction from baseline in VAS back pain score by at least 20 mm, lack of device-related serious adverse events, absence of neurologic worsening and absence of surgical re-intervention.
Time Frame: Baseline and 6 months
Population: Of 194 subjects who were eligible and signed informed consent, 10 voluntarily withdrew prior to SIJF. All data from 12 subjects at a single center were excluded due to early termination of the site. 172 subjects were treated. 168 had 6 months of follow up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sacroiliac Joint Fusion
Number analyzed (Participants) | 168
percentage of participants | 80.5 [74.0 to 85.9]

2. Secondary Outcome: Change in SI Joint Pain on Visual Analog Scale (VAS) (0-100 mm)
Description: The Visual Analog Scale (VAS) is a 100 mm line on which the subject indicates their level of pain. 0 = no pain. 100 = worst imaginable pain.
Time Frame: 24 months
Population: 148 subjects had SIJ pain scores at 24 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sacroiliac Joint Fusion
Number analyzed (Participants) | 148
units on a scale | 53.3 (27.6)

3. Secondary Outcome: Change in Back Dysfunction
Description: Oswestry Disability Index is a validated patient questionnaire aiming to assess low back pain. The computed scores can be 0% to 100%. Lower scores indicate low disability while high scores indicate high disability. There are 10 questions on the questionnaire. Each has 6 possible answers (0 points - 5 points). If the question is skipped, it's points are subtracted from the denominator. If the raw score is 30 and all 10 questions were answered, the calculation would be 30 / 50 = 60%. If one question was skipped, it would be 30 / 45 = 67%.
Time Frame: 24 months
Population: 147 of participants had ODI at 24 months post-operatively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sacroiliac Joint Fusion
Number analyzed (Participants) | 147
units on a scale | 24.5 (21.1)

4. Secondary Outcome: Change in Quality of Life
Description: Change in QOL as measured by Short Form-36 PCS and EQ-5D at post-operative visits
Time Frame: Baseline and 24 months
Population: 148 participants had QOL information at 24 months post-operatively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sacroiliac Joint Fusion
Number analyzed (Participants) | 148
units on a scale
  SF36 PCS | 8.9 (10.6)
  SF36 MCS | 10.1 (11.8)
  EQ5D TTO | .27 (.26)

5. Secondary Outcome: Ambulatory Status
Description: Percentage of population fully ambulatory at 24 months post operatively.
Time Frame: 24 months
Population: 148 participants had ambulatory status at 24 month post-operatively
Measure: Number; unit: percentage of participants
Arm/Group | Sacroiliac Joint Fusion
Number analyzed (Participants) | 148
percentage of participants | 89.2

6. Secondary Outcome: Work Status
Description: Proportion of non-working subjects who return to work
Time Frame: Basline, 24 months
Population: Participants with work status data at 24 months post-operatively who were not working due to back pain (at baseline 37.4% were not working due to back pain).
Measure: Number; unit: percentage of participants
Arm/Group | Sacroiliac Joint Fusion
Number analyzed (Participants) | 148
percentage of participants | 25.0

7. Secondary Outcome: Serious Adverse Events
Description: Occurrence of adverse events meeting the ISO14155:2011 definition of serious occurring during the procedure, at the time of hospital discharge (typically day of or next day after procedure), and at various times in late follow-up.
Time Frame: Procedure, discharge, 1,3,6,12,18 and 24 months
Population: 149 participants had 24 months of follow up post-operatively.
Measure: Number; unit: serious adverse event
Arm/Group | Sacroiliac Joint Fusion
Number analyzed (Participants) | 149
serious adverse event | 100

ADVERSE EVENTS:
Time Frame: 1 month, 3 months, 6 months, 12 months, 18 months, 24 months
Arm/Group | Sacroiliac Joint Fusion
Serious Adverse Events (participants affected / at risk) | 67/172
Other Adverse Events (participants affected / at risk) | 153/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sacroiliac Joint Fusion (N=172)
Osteoarthritis of the knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Degenerative disease - spine (Musculoskeletal and connective tissue disorders) | 12 (12)
Degenerative disease - knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Contralateral SIJ pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Ipsilateral SIJ pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Degenerative disease - Hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Wrist fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Multiple fractures and concussion MVA (Musculoskeletal and connective tissue disorders) | 1 (1)
Hammer toe (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis of the hip (Musculoskeletal and connective tissue disorders) | 2 (2)
Humerus fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertebral compression fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Ipsilateral leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Degerative disease - shoulder (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain from fractured pedicle screws (Musculoskeletal and connective tissue disorders) | 1 (2)
Dislocated shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Revision - SIJ pain (Injury, poisoning and procedural complications) | 3 (3)
Surgery site pain (Injury, poisoning and procedural complications) | 1 (1)
Revision - fusion hardware pressing on SIJF implants (Injury, poisoning and procedural complications) | 1 (1)
Revision - neuropathy post op (Injury, poisoning and procedural complications) | 2 (2)
Wound infection / irritation (Injury, poisoning and procedural complications) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Choledocholithiasis (Hepatobiliary disorders) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 2 (2)
GI bleed (Gastrointestinal disorders) | 1 (1)
Prolapsing hemorrhoids (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Morbid obesity (General disorders) | 1 (1)
Dry mouth associated tooth decay (General disorders) | 1 (1)
Suproventricular tachycardia (Cardiac disorders) | 1 (1)
Syncope with dizziness (Cardiac disorders) | 1 (1)
MI fatal (Cardiac disorders) | 1 (1)
cardiac failure septal defect (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
DVT - protein S deficient (Vascular disorders) | 1 (1)
Worsened arthrosclerosis (Vascular disorders) | 1 (1)
Pulmonary embolism with pneumonia (Vascular disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Wound infection post other surgery (Infections and infestations) | 2 (2)
Infection around pain pump (Infections and infestations) | 1 (1)
Systemic viral infection (Infections and infestations) | 1 (1)
Appendicitis (Immune system disorders) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1)
Arthritis - thumb (Immune system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypercalcemia (Endocrine disorders) | 1 (1)
Lacunar stroke (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervical cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Suicide (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sacroiliac Joint Fusion (N=172)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (37)
Foot fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Thigh pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Buttock pain (Musculoskeletal and connective tissue disorders) | 19 (20)
Cervical stenosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Cervical radiculopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Tibial plateau stress fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Ipsilateral SIJ pain (Musculoskeletal and connective tissue disorders) | 21 (24)
Degenerative disease - spine (Musculoskeletal and connective tissue disorders) | 28 (33)
Contralateral SIJ pain (Musculoskeletal and connective tissue disorders) | 18 (19)
Hip pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Knee pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Back muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Degenerative disease - hip (Musculoskeletal and connective tissue disorders) | 3 (3)
Iliotibial band syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 9 (10)
Swelling behind left knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Ankle strain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1)
hamstring tear (Musculoskeletal and connective tissue disorders) | 1 (1)
Piriformis syndrome (Musculoskeletal and connective tissue disorders) | 4 (4)
Leg, hip, groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Revision - SIJ pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Meniscal tear (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis of the wrist (Musculoskeletal and connective tissue disorders) | 1 (1)
Wrist fusion surgery implant problem (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Calf pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain due to broken lumbar fusion screws (Musculoskeletal and connective tissue disorders) | 1 (1)
Supraspinatus tear (Musculoskeletal and connective tissue disorders) | 1 (1)
Tennis elbow (Musculoskeletal and connective tissue disorders) | 2 (3)
Elbow pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteomyelitis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Radial head fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Wrist pain from punching hard object (Musculoskeletal and connective tissue disorders) | 1 (1)
AVN - hip (Musculoskeletal and connective tissue disorders) | 2 (3)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Diastasis recti (Musculoskeletal and connective tissue disorders) | 1 (1)
Numbness thigh / foot contralateral (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Calf contusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Labral tear bilaterally (Musculoskeletal and connective tissue disorders) | 1 (1)
Right L5 radicular pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Restless leg syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsened knee extension (Musculoskeletal and connective tissue disorders) | 1 (1)
Ischial tuberosity pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Knee stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Iliac crest fibrosis hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Contralateral SIJ degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Flexor sheath cyst in finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Humerus tuberosity fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar myofascial pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ankle jerk (Musculoskeletal and connective tissue disorders) | 1 (1)
Myofascial pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis of the hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Back and neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical spondylosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)
Removal of pain pump (General disorders) | 1 (1)
Spontaneous miscarriage (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Rheumatoid arthritis (Immune system disorders) | 2 (2)
Eczema (Immune system disorders) | 1 (1)
Arthritis - hands (Immune system disorders) | 1 (1)
Arthritis - ankles (Immune system disorders) | 1 (1)
Allergic rhinitis (Immune system disorders) | 1 (1)
Pruritis drug reaction (Immune system disorders) | 1 (1)
Low sensation / strength left leg (Nervous system disorders) | 1 (1)
Foot drop - left (Nervous system disorders) | 1 (1)
Ankle dorsiflexion (Nervous system disorders) | 1 (1)
Contralateral leg weakness (Nervous system disorders) | 1 (1)
Foot numbness bilateral (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 2 (2)
Fibromyalgia (Nervous system disorders) | 2 (2)
Leg numbness (Nervous system disorders) | 1 (1)
Foot numbness (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Hit head (Nervous system disorders) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1)
Right leg weakness (Nervous system disorders) | 1 (1)
Left leg sensory (Nervous system disorders) | 1 (1)
Bilateral leg neuropathic pain (Nervous system disorders) | 1 (1)
Ipsilateral thigh pain (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
L5 sensory (Nervous system disorders) | 1 (1)
Contralateral leg numbness and pain (Nervous system disorders) | 1 (1)
Cataracts (Eye disorders) | 2 (2)
Corneal abrasion (Eye disorders) | 1 (1)
Type 2 diabetes (Endocrine disorders) | 1 (1)
Hypercholesterolemia (Endocrine disorders) | 2 (2)
Osteopenia (Endocrine disorders) | 1 (1)
Diabetes mellitus (Endocrine disorders) | 1 (1)
Hypercalcemia (Endocrine disorders) | 1 (1)
Osteoporosis (Endocrine disorders) | 1 (1)
Sinusitis (Infections and infestations) | 3 (4)
Wound seroma after pain pump removal (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Infection at flu shot site (Infections and infestations) | 1 (1)
Cellulitis on leg (Infections and infestations) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Edema on leg (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Angina (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Kidney stone (Renal and urinary disorders) | 3 (3)
UTI (Renal and urinary disorders) | 5 (5)
Urinary retention (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Hiatal hernia (Gastrointestinal disorders) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 1 (1)
Bacterial gastroenteritis (Gastrointestinal disorders) | 1 (1)
Nausea (Injury, poisoning and procedural complications) | 3 (3)
Intraoperative hemorrhage 800cc (Injury, poisoning and procedural complications) | 1 (1)
Surgery site pain (Injury, poisoning and procedural complications) | 1 (1)
Right foot weakness (Injury, poisoning and procedural complications) | 1 (1)
Wound infection / irritation (Injury, poisoning and procedural complications) | 5 (5)
Revision - SIJ pain (Injury, poisoning and procedural complications) | 1 (1)
Incision site numbness (Injury, poisoning and procedural complications) | 1 (1)
Transient WBC elevation (Blood and lymphatic system disorders) | 1 (1)
Bilateral LE edema (Blood and lymphatic system disorders) | 1 (1)
Chronic lymphocytic leukemia (Blood and lymphatic system disorders) | 1 (1)
Allergic dermatitis to tape (Skin and subcutaneous tissue disorders) | 1 (2)
Finger laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Thumb laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Xanax withdrawal (Psychiatric disorders) | 1 (1)
Drug addiction (Psychiatric disorders) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1)
Abdominal aortic aneurysm (Vascular disorders) | 1 (1)
Wound bleed post cervical fusion (Vascular disorders) | 1 (1)
Numbness related to syringomyelia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ear pain - eustachian tube problem (Ear and labyrinth disorders) | 1 (1)
Cervical myelopathy (Musculoskeletal and connective tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Lack of concurrent control group undergoing non-surgical treatment and a 24-month follow up rate that was not as high as desired.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the site is that the sponsor can review results communications prior to public release and must have at least 30 days to do so.